CLINICAL TRIAL: NCT00078364
Title: Imaging Neural Mechanisms Underlying Pain Modulation
Brief Title: Pain Pathways in the Brain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 040125; 04-D-0125
Record Dates: First submitted 2004-02-23; First posted 2004-02-24 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2005-08

CONDITIONS: Healthy; Tooth Extraction
Keywords: MRI; NSAID Analgesia; Pain Mechanisms; SNP's; Acute Pain; Wisdom Teeth; Third Molar Extraction; Third Molar Impaction
MeSH Terms: conditions — Acute Pain

INTERVENTIONS:
Procedure: MRI

SUMMARY:
This study will evaluate brain pathways involved in feeling pain and pain relief following administration of pain medication. Magnetic resonance imaging (MRI) will be used to measure brain activity at sites that become more active following oral surgery and then to see if the activity changes after pain medication is administered. MRI combines a powerful magnet with an advanced computer system and radio waves to produce detailed pictures of organs and tissues. During the scan, the subject lies on a table in a narrow cylinder containing a magnetic field. He or she can speak with a staff member via an intercom system at all times during the procedure.

Healthy dental patients recruited through the NIH Clinical Research Volunteer Program may enroll in this study. Participants will undergo the following tests and procedures in two clinic visits:

Visit 1 - Sensitivity Testing

Participants are tested for sensitivity to warm and hot temperatures. A probe is applied to the skin (usually the forearm) and heated to temperatures ranging from room temperature to that of a hot cup of coffee. Participants rate the temperature using a scale ranging from "no pain" to the "worst pain imaginable" and rate the unpleasantness of the heat using a similar scale. The probe is applied up to 30 times, using random heat intensities. Participants are also asked compare the heat intensity to varying levels of sounds and to rate the magnitude of different sensations they have experienced in the past, such as the brightness of the sun and the loudness of a jet plane. A blood sample of about 2 ounces is also collected at this visit for DNA analysis to look for genes related to pain.

Visit 2 - Oral Surgery

Under local anesthetic, participants undergo extraction of their lower right wisdom tooth. After surgery, the patient is moved to the MRI scanner for brain imaging over 1-2 hours while the local anesthetic wears off. Patients may request a postoperative pain drug (Toradol) during the procedure, if needed. When the scan is complete, patients are dismissed from the clinic with additional pain medication (flurbiprofen) to use at home as directed.

DETAILED DESCRIPTION:
Functional neuroimaging provides a powerful tool for understanding how the brain may be involved in the perception of pain. It has made it possible to identify areas of the brain that are involved in the perception of experimental pain but very few studies have evaluated the sites in the brain that are activated during clinical pain and the effects of analgesic drugs. The proposed study will use the surgical removal of an impacted third molar as a model of acute clinical pain to identify sites that are activated following the offset of local anesthesia and to examine the effects of the NSAID analgesic ketorolac on attenuating sites that are activated as pain is relieved. Scans will be performed under non-pain baseline conditions, and again immediately following surgery as the local anesthetic wears off, clinical pain occurs, and following administration of the NSAID ketorolac. Differences among subjects in the amount of pain reported and brain activation will be compared to subjects' prior ratings of experimental pain and the presence of any genetic polymorphisms that are related to pain perception, inflammation, known pain pathways, or psychological factors related to pain. The findings from this research may help to reveal how pain is appreciated in the central nervous system, pharmacologically modified by NSAID analgesics and differs among individuals due to genetic factors.

ELIGIBILITY:
ELIGIBILITY CRITERIA:

Subjects will be a convenience sample selected from the pool of 500 - 700 new patients screened annually for acute pain studies. Inclusion and Exclusion criteria will be applied to result in a homogeneous population of subjects with respect to the surgical difficulty of the tooth being extracted, a single lower right third molar.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30
Dates: Start 2004-02; Study Completion 2005-08

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Dental And Craniofacial Research (NIDCR), Bethesda, Maryland, United States

REFERENCES:
- [Background] Bingel U, Quante M, Knab R, Bromm B, Weiller C, Buchel C. Subcortical structures involved in pain processing: evidence from single-trial fMRI. Pain. 2002 Sep;99(1-2):313-21. doi: 10.1016/s0304-3959(02)00157-4. PMID 12237210
- [Background] Apkarian AV, Krauss BR, Fredrickson BE, Szeverenyi NM. Imaging the pain of low back pain: functional magnetic resonance imaging in combination with monitoring subjective pain perception allows the study of clinical pain states. Neurosci Lett. 2001 Feb 16;299(1-2):57-60. doi: 10.1016/s0304-3940(01)01504-x. PMID 11166937
- [Background] Chen AC. New perspectives in EEG/MEG brain mapping and PET/fMRI neuroimaging of human pain. Int J Psychophysiol. 2001 Oct;42(2):147-59. doi: 10.1016/s0167-8760(01)00163-5. PMID 11587773